CLINICAL TRIAL: NCT07039903
Title: Bridging the Gap in the Study of Bipolar Disorder and Attention Deficit Hyperactivity Disorder: Impact of cognitiVE Reserve and funCtioning in a Newly Designed Treatment intervenTion for comORbidity (VECTOR)
Brief Title: A Novel Psychological Intervention for Adults With Bipolar Disorder and Attention Deficit Hyperactivity Disorder Comorbidity (VECTOR)
Acronym: VECTOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)041-2025; PI24/00671 and PI24/00407 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: ADHD; BD
Keywords: clinical trial; Cognitive Behavioral Therapy; Psychological treatment; Bipolar Disorder; Bipolar and Related Disorders; BD; Attention-Deficit Hyperactivity Disorder; ADHD; Functional remediation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Bipolar Disorder; Bipolar and Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VECTOR program (Experimental): The VECTOR enhancement protocol consists of 12 weekly sessions (90 minutes each of them) in a group format (8-10 individuals) with audiovisual support.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) + Functional Remediation (FR)
- Treatment as usual (TAU) (No Intervention): All participants will receive standard care in accordance with the current practice at the participating centre, respecting international recommendations for the management of their illness.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) + Functional Remediation (FR) — VECTOR will provide a newly designed intervention, based on the adaptation of two existing evidence-based and effective interventions (CBT for ADHD and FR for BD)(Corrales et al., 2024; Torrent et al., 2013).
  Arms: VECTOR program

SUMMARY:
Cognitive dysfunctions are present in Bipolar Disorder (BD) and Attention Deficit Hyperactivity Disorder (ADHD) and may negatively impact psychosocial functioning. Further, comorbid BD and ADHD (BD-ADHD) is prevalent, associated with an earlier BD onset and a less favorable prognosis. Nevertheless, there is a paucity of research dedicated to the characterization and treatment of comorbid BD-ADHD.

This study aims to develop and evaluate the effectiveness of a novel psychological group intervention (VECTOR) for adults with BD-ADHD. VECTOR integrates elements from Cognitive Behavioral Therapy (CBT) for ADHD and Functional Remediation (FR) for BD.

Eighty patients will be randomized (1:1) to receive either the VECTOR program (12 weekly group sessions) or treatment as usual (TAU).

It is expected that the VECTOR program will result in greater improvements in functioning and symptom reduction compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill DSM-5 criteria for BDI or BDII and ADHD using the Structured Clinical Interview for DSM-5 and the Conners' Adult ADHD Diagnostic Interview (CAARS)
* Aged ≥18
* Stable pharmacological treatment for at least the past three months.
* Being in full or partial remission Young Mania Rating Scale (YMRS) ≤ 10, Hamilton Depression Rating Scale (HDRS) ≤ 14) at the time of the inclusion and assessment
* ADHD rating scale≥24

Exclusion Criteria:

* Any comorbid psychiatric condition
* Diagnosis of substance abuse disorder in the past 12 months
* Intellectual disability (intelligence quotient < 70)
* Having any Central Nervous System illness, independent of primary psychiatric diagnosis, hampering neuropsychological performance
* Participation in a structured psychological intervention during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functioning Assessment Short Test (FAST) | Baseline, post-treatment (12 weeks) and 12 months
  24-item scale assessing disability in six functional domains: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, and leisure time. Assessed by a blind expert rater.
Clinical Global Impression - Severity (CGI-S) | Baseline, post-treatment (12 weeks) and 12 months
  Severity scale measuring global symptom severity. Assessed by a blind expert rater.

SECONDARY OUTCOMES:
Change in the ADHD-Rating Scale (ADHD-RS) | Baseline, post-treatment (12 weeks) and 12 months
  The ADHD-RS is an 18-items scale self-report version for assessing symptoms for ADHD DSM-IV. It consists of a subscale of inattention (IN, 9-items), another of hyperactivity/impulsivity (H / I, 9-items) and the total (TOT, 18-items). The interviewees are asked about the frequency of the symptoms over the past 6 months.
Change in the severity of ADHD symptoms | Baseline, post-treatment (12 weeks) and 12 months
  Assessed by Connors' Adult ADHD Rating Scales Self-report form (CAARS-S:L), a self-report questionnaire evaluating the severity of ADHD symptoms across multiple domains, including inattention and hyperactivity/impulsivity.
Change in the severity of ADHD symptoms | Baseline, post-treatment (12 weeks) and 12 months
  Assessed by Connors' Adult ADHD Rating Scales Observer form (CAARS-O-L), an observer-rated questionnaire assessing ADHD symptom severity based on third-party observation, covering the same symptom domains as the self-report version.
Change in the Hamilton Depression | Baseline, post-treatment (12 weeks) and 12 months
  Each item is rated on either a 3-point or 5-point Likert-type scale, depending on the symptom being assessed, with higher scores indicating greater severity of depression. The total score for the HDRS-17 ranges from 0 to 52. Common domains evaluated include mood, guilt, suicide ideation, insomnia, anxiety, psychomotor changes, and somatic symptoms.
Change in the Young Mania Rating Scale (YMRS) | Baseline, post-treatment (12 weeks) and 12 months
  11-item clinician-rated scale used to assess manic symptoms such as elevated mood, increased motor activity, sleep disturbance, irritability, and thought disorder. Higher scores reflect more severe manic symptoms. Assessed by a blind expert rater.
Change in attention - Trail Making Test Part A (TMT-A) | Baseline, post-treatment (12 weeks) and 12 months
  TMT-A assesses processing speed and visual attention. Participants are asked to connect numbered circles in sequence as quickly as possible. Completion time is the outcome measure; shorter times indicate better performance.
Change in cognitive flexibility - Trail Making Test Part B (TMT-B) | Baseline, post-treatment (12 weeks) and 12 months
  TMT-B assesses cognitive flexibility, task-switching, and executive control. Participants alternate between numbers and letters in sequence (e.g., 1-A-2-B...). Completion time is recorded, with shorter times indicating better performance.
Change in sustained attention - Conners' Continuous Performance Test (CPT) | Baseline, post-treatment (12 weeks) and 12 months
  The CPT is a computerized test that measures sustained attention and impulsivity by recording responses to a series of visual stimuli. Key outcomes include omission errors, commission errors, and reaction time variability.
Change in executive function - Wisconsin Card Sorting Test (WCST) | Baseline, post-treatment (12 weeks) and 12 months
  The WCST measures cognitive flexibility and executive functioning. Participants must match cards according to varying rules. Key outcomes include number of categories completed and perseverative errors.
Change in inhibitory control - Stroop Test | Baseline, post-treatment (12 weeks) and 12 months
  The Stroop Color-Word Test evaluates selective attention and inhibitory control by measuring the ability to name the color of the ink rather than reading the printed word. Interference score is commonly used.
Change in verbal fluency - Phonemic and Semantic Fluency (PMR) | Baseline, post-treatment (12 weeks) and 12 months
  The Verbal Fluency Test assesses executive control and language by requiring the participant to generate as many words as possible starting with a letter (phonemic) or within a category (semantic) in a limited time.

OTHER OUTCOMES:
CSQ-8 | 12 weeks (post)
  Client Satisfaction Questionnaire-8 (self-report) - in order to evaluate the treatment satisfaction
Working Alliance Inventory | 12 weeks (post)
  The Working Alliance Inventory (WAI) is a self-report questionnaire designed to assess the quality of the therapeutic relationship. It evaluates three key components: agreement on therapeutic goals, agreement on tasks, and the emotional bond between therapist and patient. Higher scores indicate a stronger working alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona and Vall d'Hebron University Hospital, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) due to ethical and legal constraints related to data privacy and participant confidentiality, in accordance with applicable regulations and institutional policies.

REFERENCES:
- [Background] Torrent C, Bonnin Cdel M, Martinez-Aran A, Valle J, Amann BL, Gonzalez-Pinto A, Crespo JM, Ibanez A, Garcia-Portilla MP, Tabares-Seisdedos R, Arango C, Colom F, Sole B, Pacchiarotti I, Rosa AR, Ayuso-Mateos JL, Anaya C, Fernandez P, Landin-Romero R, Alonso-Lana S, Ortiz-Gil J, Segura B, Barbeito S, Vega P, Fernandez M, Ugarte A, Subira M, Cerrillo E, Custal N, Menchon JM, Saiz-Ruiz J, Rodao JM, Isella S, Alegria A, Al-Halabi S, Bobes J, Galvan G, Saiz PA, Balanza-Martinez V, Selva G, Fuentes-Dura I, Correa P, Mayoral M, Chiclana G, Merchan-Naranjo J, Rapado-Castro M, Salamero M, Vieta E. Efficacy of functional remediation in bipolar disorder: a multicenter randomized controlled study. Am J Psychiatry. 2013 Aug;170(8):852-9. doi: 10.1176/appi.ajp.2012.12070971. PMID 23511717
- [Background] Corrales M, Garcia-Gonzalez S, Richarte V, Fadeuilhe C, Daigre C, Garcia-Gea E, Ramos-Quiroga JA. Long-term efficacy of a new 6-session cognitive behavioral therapy for adults with attention-deficit/hyperactivity disorder: A randomized, controlled clinical trial. Psychiatry Res. 2024 Jan;331:115642. doi: 10.1016/j.psychres.2023.115642. Epub 2023 Nov 27. PMID 38103281
- [Background] Amoretti S, De Prisco M, Clougher D, Garriga M, Corrales M, Fadeuilhe C, Forte MF, Martinez-Aran A, Oliva V, Parramon-Puig G, Richarte V, Amann BL, Oliva F, Ruiz A, Sole B, Valenti M, Crespin JJ, Arteaga-Henriquez G, Vieta E, Ramos-Quiroga JA, Torrent C. Neurocognitive and psychosocial functioning profiles in bipolar disorder and comorbid attention deficit hyperactivity disorder: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2025 Apr;171:106081. doi: 10.1016/j.neubiorev.2025.106081. Epub 2025 Feb 26. PMID 40015388